CLINICAL TRIAL: NCT01377961
Title: Effect of Lycopene and Isoflavones on Glucose Metabolism
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: FDA needs more information from the manufacturing company of the supplements.
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10-065
Record Dates: First submitted 2011-03-30; First posted 2011-06-22 (Estimated); Last update posted 2015-06-26 (Estimated); Status verified 2015-06

CONDITIONS: Metabolic Syndrome; Diabetes Mellitus, Non-Insulin-Dependent
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus, Type 2 | interventions — Isoflavones; Dietary Supplements; Mass Screening; Glucose Tolerance Test; Blood Pressure; Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm1: Metabolic Syndrome Volunteers (Active Comparator)
  Interventions: Drug: Randomized pills either containing combination of lycopene and isoflavones (dietary supplements) or Placebo to be taken for 12 weeks; Other: Screening; Other: OGTT; Other: Anthropometrics and Blood pressure; Other: Blood Drawing
- Arm 2:Previously Diagnosed diabetic patients (Active Comparator)
  Interventions: Drug: Randomized pills either containing combination of lycopene and isoflavones (dietary supplements) or Placebo to be taken for 12 weeks; Other: Screening; Other: Anthropometrics and Blood pressure; Other: Blood Drawing

INTERVENTIONS:
Drug: Randomized pills either containing combination of lycopene and isoflavones (dietary supplements) or Placebo to be taken for 12 weeks — After the screening and OGTT, the treatment group each subject will be in is decided by randomization. Neither subject nor the researchers will be allowed to choose which group a subject is assigned to. A single patient/subject cannot be assigned more than 1 allocation number. Each subject will be assigned randomly (like drawing straws) to receive either on the pills containing the combination of 6mg lycopene and 50mg isoflavones or placebo. Each subject has a 1 in 2 chance of receiving one of these treatments.
  The subject are advised to take one capsule of Laflavon/Placebo by mouth daily for 12 weeks.
Other: Screening — Volunteer will be screened as an out patient with a history, physical examination, baseline fasting plasma glucose or A1C, creatinine, AST/ALT, TSH. We may utilize the lab results of the subject available upto 3months prior to the consent date. Pregnancy tests will be performed for female candidates. Information of the level of physical activity, diet, supplements and medications will be obtained.
Other: OGTT — OGTT will be done after the screening at Baseline and at the completion of the 12 weeks of taking the supplements by the subject.
  Arms: Arm1: Metabolic Syndrome Volunteers
Other: Anthropometrics and Blood pressure — Measurements of height, weight, hip, waist and Blood Pressure are done before and after 12 weeks of taking the supplements.
Other: Screening — Volunteer will be screened as an out patient with a history, physical examination, baseline fasting plasma glucose or A1C, creatinine, AST/ALT, TSH. We may utilize the lab results of the subject available upto 3months prior to the consent date. Pregnancy tests will be performed for female candidates. Information of the level of physical activity, diet, supplements and medications will be obtained.
  Arms: Arm 2:Previously Diagnosed diabetic patients
Other: Blood Drawing — The blood will be drawn at the baseline and at the completion of the 12 weeks of taking the capsules of laflavon /placebo.

SUMMARY:
Type 2 diabetes mellitus (DM2) is a growing social health problem world-wide, in particular with respect to its contribution to cardiovascular disease. The progressive increase in prevalence of DM2 has reached epidemic proportion and is a major cause of morbidity and mortality in all populations around the world. Conventional stepwise treatment of DM2 generally focuses on controlling blood glucose concentration. However, the risk for side-effects associated with the use of pharmacological intervention often delays initiation of therapy, with the potential implication on worsening morbidity and mortality from complications. On the other hand, non-pharmacological intervention in the form of dietary restrictions, exercise and weight loss, is safe but often difficult to accomplish. The availability of nutrients that affect glucose and lipid metabolism would provide an important practical tool to establish early intervention in newly diagnosed DM2 and perhaps even in patients who are only "at risk" for DM2. The investigators have recently obtained preliminary data on beneficial effects of combined supplementation of lycopene and isoflavones on glucose metabolism of normoglycemic volunteers with insulin resistance. This clinical trial will explore the role of isoflavones and lycopene dietary supplementation in the improvement of glucose metabolism of patients at increased risk or with established but mild DM2. The overall hypothesis is that supplementation of laflavon, provided as a new formulation that increases bioavailability of the individual components (Laflavon CamMedica contains 7 mg of Lycopene and 50 mg of Soy Isoflavones), determines improvement in glucose tolerance and insulin resistance of patients with the metabolic syndrome and also reduces HbA1c in patients with mild DM2.

ELIGIBILITY:
Study group 1( arm 1 ::metabolic syndrome group).

Inclusion criteria:

* Age 18-75 years
* Metabolic Syndrome (IDF criteria)
* Stable dose of medications for > 90 days

Exclusion criteria:

* Pharmacological therapy for diabetes
* Flood allergies, especially to Whey protein, soy or tomato.
* Pregnancy

Study group 2( Arm 2:: Diabetes mellitus patients group).

Inclusion criteria:

* 18-75 years of age
* Type 2 diabetes (diagnosed with ADA criteria: fasting plasma glucose > 125 mg/dL)
* Stable dose of medications for > 90 days
* Patients on diet/exercise, metformin, DD4 inhibitors (sitagliptin and saxagliptin) and /or sulphonylurea for > 90 days

Exclusion criteria:

* HbA1c above 9.5% or below 7.5% in last 3 months
* TZD therapy for diabetes
* Insulin therapy for diabetes
* Flood allergies, especially to Whey protein, soy or tomato
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-09; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Insulin Resistance | 12 weeks
  For Arm 1:Assessment of the Changes in the insulin resistance from baseline to 12 weeks.
A1C | 12 weeks
  For Arm 2:Assessment of the Changes in the A1C from baseline to 12 weeks.

SECONDARY OUTCOMES:
For Arm 1 :AUCglucose | 12 weeks
  For Arm 1: Changes of AUCglucose from baseline to 12 weeks.
For Arm1 and Arm 2: The secondary outcome measure are Plasma Lipids concentrations | 12 weeks
  For Arm 2: Changes in the Plasma Lipids concentrations,BMI,Plasma lycopene and isoflavones, EPCs count and function, Chlamydia Trachomatis titers in serum from baseline to 12 weeks.
For Arm 1 :AUCglucose,Plasma Lipids concentrations,BMI,Plasma lycopene and isoflavones concentration,EPCs count and function,Chlamydia Trachomatis titers in serum | 12 weeks
  For Arm 1: Changes of AUCglucose,Plasma Lipids concentrations,BMI,Plasma lycopene and isoflavones,EPCs count and function,Chlamydia Trachomatis titers in serum from baseline to 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Abate, MD, Principal Investigator — UTMB
Locations (2):
- United States (2):
  - Internal Medicine, Galveston, Texas
  - Stark Diabetes Center Clinic, Galveston, Texas